CLINICAL TRIAL: NCT05229484
Title: Effects of an Integrated Multimodal Lifestyle Intervention for Management of Violence Through Regulation of Serum Lipid Profile in Schizophrenia: A Randomized Controlled Trial
Brief Title: Effects of an Integrated Multimodal Lifestyle Intervention for Management of Violence in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I-Shou University (Other)
Responsible Party: Principal Investigator, Mei-Chi Hsu, Professor, I-Shou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IShouU-cholesterol I
Record Dates: First submitted 2022-01-06; First posted 2022-02-08 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
Keywords: Lifestyle Intervention; Management of Violence; Lipid Profile
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: an integrated multimodal lifestyle intervention (MLifeI) (Experimental): The MLifeI program focused on the roles of health responsibility, review of lipid profile, complications of imbalanced lipid profile, lipid management and nutritional education.
  Interventions: Other: an integrated multimodal lifestyle intervention (MLifeI)
- Control group (No Intervention): The control group is the Treatment as Usual (TAU).

INTERVENTIONS:
Other: an integrated multimodal lifestyle intervention (MLifeI) — The MLifeI program focused on the roles of health responsibility, review of lipid profile, complications of imbalanced lipid profile, lipid management and nutritional education.
  Arms: Intervention Group: an integrated multimodal lifestyle intervention (MLifeI)

SUMMARY:
Total cholesterol levels and other lipids are associated with violence in psychiatric patients. There is a paucity of studies on preventive interventions. In this study, an integrated multimodal lifestyle intervention (MLifeI) for management of repetitive violence in schizophrenia is proposed. A controlled clinical trial was carried out to evaluate the effects of MLifeI on management of repetitive violence through regulation of serum lipids, TC in particular, to the recommended levels in schizophrenia. The investigators examined whether the MLifeI could: 1. regulate or balance lipid profiles; 2. reduce violence risk; 3. improve impulsivity; and 4. improve general cognitive functioning.

DETAILED DESCRIPTION:
Total cholesterol levels and other lipids are associated with violence in psychiatric patients. There is a paucity of studies on preventive interventions. In this study, an integrated multimodal lifestyle intervention (MLifeI) for management of repetitive violence in schizophrenia is proposed. A controlled clinical trial was carried out to evaluate the effects of MLifeI on management of repetitive violence through regulation of serum lipids, TC in particular, to the recommended levels in schizophrenia. The investigators examined whether the MLifeI could: 1. regulate or balance lipid profiles; 2. reduce violence risk; 3. improve impulsivity; and 4. improve general cognitive functioning. The multimodal lifestyle intervention included psychoeducation, lifestyle modification and health promotion and exercise. Outcome measures comprised lipid profiles, body mass index and violence-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia for more than 2 years
* Psychiatrically hospitalized
* Repetitive violence within one year
* Ambulatory
* Having basic literacy
* More than 20 years old
* Less than 65 years old

Exclusion Criteria:

* Clinical psychiatric diagnosis other than schizophrenia
* Physical co-morbidity or life-threatening illnesses that may impact on lipid homeostasis
* dietary restrictions for physical condition
* pregnancy
* reported disabilities
* impairments or health illness/problems that significantly limited their ability to perform the intervention such as severe arthritis, uncorrected visual or hearing impairments, developmental disability, or signs of intellectual disability.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Weight in kilograms | Change of weight from baseline and 6 months (3-month follow-up)
  Clinical Assessment: weight.
Height in meters | Change of weight from baseline and 6 months (3-month follow-up)
  Clinical Assessment: height.
Body Mass Index (BMI) | Change of weight from baseline and 6 months (3-month follow-up)
  Clinical Assessment: Body Mass Index; Weight and height will be combined to report BMI in kg/m^2. The World Health Organisation defines an adult who has a BMI between 25 and 29.9 as overweight - an adult who has a BMI of 30 or higher is considered obese - a BMI below 18.5 is considered underweight, and between 18.5 to 24.9 a healthy weight.
Routine test in the ward of total cholesterol, triglyceride, low-density lipoprotein and high-density lipoprotein (Change is being assessed, mg/dL) | Change of violence risk from baseline (T1) and 6 months (T3, 3-month follow-up)
  Lipid profiles. Assessment of serum metabolites.
Violence Risk Screening (Change is being assessed) | Change of violence risk from baseline (T1), 3 months (T2, end of treatment), and 6 months (T3, 3-month follow-up)
  Questionnaires of violence. A higher score indicates a higher violence risk.
Attribution Questionnaire (Change is being assessed) | Change of violence risk from baseline (T1), 3 months (T2, end of treatment), and 6 months (T3, 3-month follow-up)
  Questionnaires of violence attributions. The Attribution Questionnair was applied to measure the participant's internal/external attributions about the causality and likelihood of violence and responsibility for changing the behavior. The measure was rated on a continuum scale from 1 (e.g., not at all likely; not at all able, etc.) to 7 (e.g., totally due to me; totally likely; totally able, etc.).
Modified Overt Aggression Scale (Change is being assessed) | Change of violence risk from baseline (T1), 3 months (T2, end of treatment), and 6 months (T3, 3-month follow-up)
  Questionnaires of aggression frequency.
Buss-Perry Aggression Questionnaire (Change is being assessed) | Change of violence risk from baseline (T1), 3 months (T2, end of treatment), and 6 months (T3, 3-month follow-up)
  Questionnaires of violence/aggression. The higher the score is, the higher the participant has the violent behavior.
Barratt Impulsiveness Scale (Change is being assessed) | Change of violence risk from baseline (T1), 3 months (T2, end of treatment), and 6 months (T3, 3-month follow-up)
  Questionnaires of impulsivity. The score ranged from 1 (rarely/never) to 4 (almost always/always). The higher the scores indicates the greater the impulsivity.
Mini-Mental State Examination (Change is being assessed) | Change of violence risk from baseline (T1), 3 months (T2, end of treatment), and 6 months (T3, 3-month follow-up)
  Questionnaires of cognitive functioning. The MMSE ranged from 0 to 30, where higher scores indicate better cognitive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chi Hsu, Ph.D, Principal Investigator — I-Shou University
Locations (1):
- I-Shou University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No